CLINICAL TRIAL: NCT06961734
Title: Effects of a Fatmax Exercise Intervention During Different Menstrual Cycle Phases on Fat Metabolism and Body Composition in Normal Weight Obese Women
Brief Title: Fatmax Exercise in Menstrual Phases: Effects on Fat Metabolism & Body Composition in NWO Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EFEIDDMCPFMBCNWOW
Record Dates: First submitted 2025-04-20; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2023-02

CONDITIONS: Fat Metabolism
Keywords: aerobic exercise; menstrual cycle phase; normal weight obesity; lipid metabolism
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- follicular group (Active Comparator)
  Interventions: Behavioral: follicular group
- luteal group (Active Comparator)
  Interventions: Behavioral: luteal group
- Control group (Active Comparator)
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: follicular group — Exercised at Fatmax intensity four times per week and plus three additional exercise during the late follicular phase of each cycle.
  Arms: follicular group
Behavioral: luteal group — Exercised at Fatmax intensity four times per week and plus three additional exercise during the mid- luteal phase of each cycle.
  Arms: luteal group
Behavioral: Control group — Exercised at Fatmax intensity four times per week.
  Arms: Control group

SUMMARY:
Effects of a Fatmax exercise intervention during different menstrual phases on fat metabolism and body composition in NWO women

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 3 arms (control group , follicular group and luteal group), in which a pre-treatment-posttest design has been used.

ELIGIBILITY:
Inclusion Criteria:

* Criteria: Inclusion Criteria:
* Female, aged between 18 and 30 years old;
* BMI between 18.5 and 24.9 kg/m2 with a BF% > 30% (normal weight obesity determination criteria);
* Regular menstrual cycles for at least 3 months;
* No use of oral contraceptives for at least 6 months before the experiment;
* Non-smoker and non-alcohol abuser.

Exclusion Criteria:

* The presence of CVD;
* A diagnosis of cancer, pulmonary diseases, or other conditions that prevent participation in exercise;
* The use of medications affecting body composition or metabolism.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Lipid profile | 8 weeks
  The changes of high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, total cholesterol, and triglyceride before and after intervention.
Body Fat Mass | 8 weeks
  Body fat mass (kg) will be assessed using dual-energy X-ray absorptiometry (DXA) scans. The change of body fat mass before and after intervention.
Percentage of Body Fat | 8 weeks
  The change of percentage of body fat before and after intervention.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 8 weeks
  Changes in Body mass index before and after Intervention. Body mass index is calculated from the formula, Weight (kg) / Height2 (m2), its unit is kg/m2.
Waist Circumference | 8 weeks
  The change of waist circumference before and after intervention.
Hip Circumference | 8 weeks
  The change of hip circumference before and after intervention.
Apolipoprotein A-I (g/L) | 8 weeks
  The change in apolipoprotein A-I levels before and after the intervention.
Apolipoprotein B (g/L) | 8 weeks
  The change in apolipoprotein B levels before and after the intervention.
Maximal Oxygen uptake (VO2max) | 8 weeks
  Changes in Maximal Oxygen uptake before and after Intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: No